CLINICAL TRIAL: NCT02524483
Title: Influence of Exercise on the Mobility and Balance of Individuals With Multiple Sclerosis Influence of High-Dosage Physical Therapy on the Balance and Mobility of Individuals With Multiple Sclerosis
Brief Title: Influence of Exercise on the Mobility and Balance of Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0467-14-EP
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

ARMS (2):
- Therapeutic Challenge Group (Experimental): The Therapeutic Challenge Group will complete the Therapeutic Challenge Program twice a day, five days each week for 6 weeks.
  Interventions: Behavioral: Therapeutic Challenge Program
- Therapeutic Exercise Group (Active Comparator): The Therapeutic Exercise Group will complete the Therapeutic Exercise Program twice a day, five days each week for 6 weeks.
  Interventions: Behavioral: Therapeutic Exercise Program

INTERVENTIONS:
Behavioral: Therapeutic Challenge Program — The Therapeutic Challenge Program will consist of a 5 minute warm-up, 20 minutes of challenging balance training, and 20 minutes of challenging treadmill and overground walking.
  Arms: Therapeutic Challenge Group
Behavioral: Therapeutic Exercise Program — The Therapeutic Exercise Program will consist of 15 minutes of strength training and flexibility exercises, 15 minutes of balance exercises, and 15 minutes of treadmill walking.
  Arms: Therapeutic Exercise Group

SUMMARY:
Outcomes from the investigators' recent investigation suggested that a high dosage of challenging physical therapy exercises can result in clinically improvements in the postural balance and walking speed of individuals with MS.

This investigation will evaluate mobility and postural balance improvements in individuals with MS who participate in a therapeutic protocol consisting of activity based exercises, and in individuals with MS that participate in challenging physical therapy protocol.

DETAILED DESCRIPTION:
Background: Outcomes from the investigators' recent exploratory investigation suggested that a high dosage of challenging physical therapy exercises can result in clinically relevant improvements in the postural balance and walking speed of individuals with MS.

Objective: The investigators anticipated that the promising results were due to the novel challenging postural balance and mobility exercises. The purpose of this investigation was to test this notion by evaluating the mobility and postural balance improvements that could be achieved in a cohort of individuals with MS who participated in a therapeutic protocol that consisted of activity based exercises, and a cohort of individuals with MS that participated in the challenging physical therapy protocol.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of multiple sclerosis
* Kurtzke Expanded Disability Status of 3.0 - 6.5
* Able to walk on a treadmill at a minimum of 0.5 miles per hour while holding onto handrails
* Cognitively and emotionally competent
* A Mini-Mental State Examination score > 21
* Composite score on the computerized Sensory Organization Test of < 70

Exclusion Criteria:

* Documented MS-related relapse in the previous 6 months
* Major MS-specific medication changes within the previous 3 months
* Presence of another major co-morbidity such as neurological disorders, uncontrolled pain, hypertension, and diabetes

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in Balance Using the Sensory Organization Test | Baseline and 6 weeks
  The Sensory Organization Test consists of six different conditions that measure each subject's ability to integrate visual, somatosensory, and vestibular feedback to reduce the overall amount of postural sway and improve balance.
Changes in Walking Velocity, Step Lengths, Step Widths, and Cadence | Baseline and 6 weeks
  The changes in walking velocity, step lengths, step widths, and cadence will be quantified using a GaitRITE digital mat.

SECONDARY OUTCOMES:
Changes in Endurance using the 6-Minute Walk | Baseline and 6 weeks
  The changes in endurance will be evaluated using the total distance walking during a 6 minute time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Max J Kurz, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Monroe-Meyer Institute, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Davies BL, Arpin DJ, Liu M, Reelfs H, Volkman KG, Healey K, Zabad R, Kurz MJ. Two Different Types of High-Frequency Physical Therapy Promote Improvements in the Balance and Mobility of Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Dec;97(12):2095-2101.e3. doi: 10.1016/j.apmr.2016.05.024. Epub 2016 Jul 1. PMID 27373745